CLINICAL TRIAL: NCT04981704
Title: A Three-Part, Open-Label, Fixed-Sequence Study to Evaluate the Effect of Multiple Doses of Itraconazole, Phenytoin, and Paroxetine on the Single-Dose Pharmacokinetics of Poziotinib in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Itraconazole, Phenytoin, and Paroxetine on the Single-Dose Pharmacokinetics of Poziotinib in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: SPI-POZ-103
Record Dates: First submitted 2021-06-23; First posted 2021-07-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — HM781-36B; Itraconazole; Phenytoin; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Itraconazole/Poziotinib Drug-drug interaction (DDI) (Experimental): On Day 1 of Treatment period 1, a single oral dose of 8 milligrams (mg) poziotinib will be administered. On Day 1 of Treatment Period 2, 200 mg itraconazole oral solution will be administered twice a day (BID) followed by 200 mg itraconazole oral solution once daily (QD) for 7 consecutive days (Day 2 to Day 8) with a single oral dose of 8 mg poziotinib coadministered on Day 4.
  Interventions: Drug: Poziotinib; Drug: Itraconazole
- Part 2: Phenytoin/Poziotinib DDI (Experimental): On Day 1 of Treatment period 1, a single oral dose of 16 mg poziotinib will be administered. In treatment period 2, an oral dose of 100 mg phenytoin will be administered three times daily (TID) for 17 consecutive days (Day 1 to Day 17) with a single oral dose of 16 mg poziotinib coadministered on Day 14.
  Interventions: Drug: Poziotinib; Drug: Phenytoin
- Part 3: Paroxetine/Poziotinib DDI (Experimental): On Day 1 of Treatment Period 1, a single oral dose of 8 mg poziotinib will be administered. On Day 1 and Day 2 of Treatment Period 2, an oral dose of 20 mg paroxetine will be administered BID followed by 20 mg paroxetine QD for 9 consecutive days (Day 3 to Day 11) with a single oral dose of 8 mg poziotinib coadministered on Day 7.
  Interventions: Drug: Poziotinib; Drug: Paroxetine

INTERVENTIONS:
Drug: Poziotinib — Poziotinib Tablets
Drug: Itraconazole — Itraconazole Oral solution
  Arms: Part 1: Itraconazole/Poziotinib Drug-drug interaction (DDI)
Drug: Phenytoin — Phenytoin Capsules
  Arms: Part 2: Phenytoin/Poziotinib DDI
Drug: Paroxetine — Paroxetine Tablets
  Other Names: Paxil ®
  Arms: Part 3: Paroxetine/Poziotinib DDI

SUMMARY:
The purpose of the study is to evaluate the effect of multiple-doses of itraconazole, phenytoin and paroxetine on the single-dose pharmacokinetics (PK) of poziotinib in healthy adult participants.

DETAILED DESCRIPTION:
This is a three-part study. Participants will be enrolled in Part 1 (Effects of Itraconazole), Part 2 (Effects of Phenytoin), or Part 3 (Effects of Paroxetine) on the Pharmacokinetics of Poziotinib. Each part will be an open-label, fixed-sequence, 2-period study and may be conducted concurrently. For each study part, participants will be housed on Day -1 of Treatment Period 1 in the Clinical Research Unit (CRU) and will remain confined in the CRU until after the last scheduled blood draw and/or study procedures in Treatment Period 2. In each part, there will be a washout period of at least 8 days between poziotinib doses.

A total of 75 (25 in each part) healthy, adult male and female participants will be enrolled targeting a female/male ratio greater than or equal to (≥) 1:3 in each study part.

In part 1, CYP2D6 extensive metabolizers will be primarily enrolled with a goal of enrolling at least 2 CYP2D6 poor metabolizers. In Parts 2 and 3, only CYP2D6 extensive metabolizers will be enrolled. In Part 2, CYP2C9 and CYP2C19 poor metabolizers will be excluded.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy, adult, male or female (of non-childbearing potential only), 18-55 years of age.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilogram per meter square (kg/m^2) at screening, and a minimum weight of 50.0 kg and a maximum weight of 100.0 kg at screening.
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study.
* Medically healthy with no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs, and laboratory evaluations.
* Female must be of non-childbearing potential only and must have undergone a sterilization procedure at least 6 months prior to the first dosing, or
* Postmenopausal women should have amenorrhea for at least 1 year prior to the first dosing.
* A non-vasectomized male participant must agree to use a highly effective method of birth control with female partners of childbearing potential or with pregnant partners during the study and for 120 days following last dosing.
* Able to comprehend and willing to sign an Informed Consent Form (ICF) and abide by the clinical protocol, study procedures, and restrictions.
* For Part 1 only: Participant must be a CYP2D6 extensive metabolizer or CYP2D6 poor metabolizer as determined by a valid genotyping method.
* For Part 2 only: Participant must not be a CYP2C9 and CYP2C19 poor metabolizer as determined by a valid genotyping method and must be a CYP2D6 extensive metabolizer as determined by a valid genotyping method.
* For Part 3 only: Participant must be a CYP2D6 extensive metabolizer as determined by a valid genotyping method.

Key Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the PI (or designee).
* History of a developing or established acute event or infection in the prior 2 weeks to screening.
* History of significant hypersensitivity, or idiosyncratic reaction to poziotinib, itraconazole, phenytoin, paroxetine, or related drugs, food, or other substances.
* Any surgical or medical condition within 6 months prior to first dosing that may potentially alter absorption, distribution, metabolism or excretion of the study drugs, in the opinion of the PI (or designee).
* History or presence of alcoholism or drug/chemical abuse within 2 years prior to check-in.
* Female participants with a positive pregnancy test result or lactating.
* Positive urine drug or alcohol test results at screening or check-in.
* Positive hepatitis panel (hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) and/or positive human immunodeficiency virus (HIV) test at screening. Automatic reflex Differential and ribonucleic acid testing will be conducted in the event of a reactive antibody/antigen screen.
* Seated blood pressure is less than 90/40 millimetre of mercury (mmHg) or greater than 140/90 mmHg at screening.
* Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
* QT interval with Fridericia's correction (QTcF) interval is >450 millisecond (msec) (males) or >470 msec (females).
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dosing and throughout the study. Hormone replacement therapy will not be allowed.
  * Any drugs known to be inhibitors and/or inducers of CYP3A, CYP2D6, CYP2C9, or CYP2C19 enzymes; and/or P-gp; and/or gastric acid reducing agents (proton-pump inhibitors, H2-receptor antagonists, antacids) for 28 days prior to the first dosing and throughout the study (except those required as part of the study).
* Has a coagulation test (i.e., prothrombin time and activated partial thromboplastin time) outside of normal ranges at screening or at check-in.
* Has platelet, hemoglobin, or hematocrit that are below the lower limit of normal at screening or at check-in.
* Has alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin that are greater than the upper limit of normal at screening or at check-in.
* Estimated creatinine clearance <90 milliliter per minute (mL/min) at screening.
* Participation in another clinical study within 30 days prior to the first dosing.
* Prior exposure to poziotinib.
* For Part 1 Only:History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and as confirmed by the Sponsor:

  * Ventricular dysfunction or risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, family history of Long QT Syndrome).
  * Uncorrected hypokalemia (potassium levels < 3.7) and/or hypomagnesemia (magnesium levels < 1.9).
  * Myasthenia gravis.
* For Part 2 Only: History of seizure (excluding simple febrile seizure), epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions which the Investigator considers to be clinically significant.
* Is at suicidal risk in the opinion of the PI as per the following criteria:

  * Any suicidal attempts within 12 months prior to screening.
  * any suicidal intent including a plan or C-SSRS answer of "YES" on suicidal ideation currently or within 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of Poziotinib and Metabolites (M1 and M2) Following Poziotinib Administrations With and Without Itraconazole [Part 1], Phenytoin [Part 2], or Paroxetine [Part 3] | Part 1 and Part 3, predose and up to 120 hours postdose; Part 2, predose and up to 96 hours postdose
Maximum Observed Concentration (Cmax) of Poziotinib and Metabolites (M1 and M2) Following Poziotinib Administration With and Without Itraconazole [Part 1], Phenytoin [Part 2], or Paroxetine [Part 3] | Part 1 and Part 3, predose and up to 120 hours postdose; Part 2, predose and up to 96 hours postdose
Apparent Clearance (CL/F) of Poziotinib Following Poziotinib Administration With and Without Itraconazole [Part 1], Phenytoin [Part 2], or Paroxetine [Part 3] | Part 1 and Part 3, predose and up to 120 hours postdose; Part 2, predose and up to 96 hours postdose
Time to Maximum Observed Concentration (Tmax) for Poziotinib and Metabolites (M1 and M2) Following Poziotinib Administration With and Without Itraconazole [Part 1], Phenytoin [Part 2], or Paroxetine [Part 3] | Part 1 and Part 3, predose and up to 120 hours postdose; Part 2, predose and up to 96 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening, and up to 14 days post last dose of Poziotinib
Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters From Baseline | Screening, and up to 14 days post last dose of Poziotinib
  Clinical laboratory parameters include tests of hematology, chemistry, coagulation, and urinalysis.
Number of Participants With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG) Findings From Baseline | Screening, and up to 14 days post last dose of Poziotinib
Number of Participants With Clinically Significant Changes in Vital Signs From Baseline | Screening, and up to 14 days post last dose of Poziotinib
  Vital signs include body temperature, respiratory rate, blood pressure, and heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (1):
- Celerion, Phoenix clinical facility, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No